CLINICAL TRIAL: NCT02845778
Title: Pharmacokinetics of Melatonin Niosomes Oral Gel in Healthy Volunteers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Supawan Laohasiriwong, Department of Otorhinolaryngology, Faculty of Medicine, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: IN58358
Record Dates: First submitted 2016-07-24; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Pharmacokinetics of Melatonin
Keywords: melatonin; pharmacokinetics
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- melatonin niosomes oral gel 2.5 mg (Experimental): apply onto oral mucosa as single use
  Interventions: Drug: Melatonin
- melatonin niosomes oral gel 5 mg (Experimental): apply onto oral mucosa as single use
  Interventions: Drug: Melatonin
- melatonin niosomes oral gel 10 mg (Experimental): apply onto oral mucosa as single use
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Each sachet contains 0.5 g
  Other Names: Melatonin niosomes oral gel 5 mg/g; Melatonin niosomes oral gel 10 mg/g; Melatonin niosomes oral gel 20 mg/g

SUMMARY:
Melatonin is an endogenous hormone. It is able to promote nighttime sleeping and could induce sleep at daytime in adult and children with the nonpainful diagnostic procedure. However, previous formulation had problems of unstability of product and low oral bioavailability. Melatonin niosomes oral gels are formulated in order to overcome the problem of drug absorption and stability. This study is a randomized, double-blind, three phase crossover design in 15 male volunteers. Melatonin niosomes oral gel will be applied at doses 2.5, 5, and 10 mg with 7 days washout for each period. The pharmacokinetics data, sleep induction effect, and adverse event will be determined.

DETAILED DESCRIPTION:
This study will determine the pharmacokinetics, sleep induction effect, and adverse event after apply melatonin niosomes (MN) oral gel 2.5, 5, and 10 mg per dose in 15 male healthy volunteers. The pharmacokinetic parameters include maximum plasma concentration (Cmax), area under the curve (AUC), time to peak concentration (Tmax), elimination half-life (t1/2). Sleep induction will be determined as sleep onset and duration after use MN oral gels using actigraph and behavior observation. A polysomnography using electrode placement derive from multiple sleep latency test (MSLT) protocol will be used in some subjects. Adverse event will be evaluated by investigator.

ELIGIBILITY:
Inclusion Criteria:

* male
* age 18-30 years
* body mass index 18.5-25 kg/m2
* general good health and no underlying disease by physical examination and laboratory testing (blood urea nitrogen, creatinine, bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, complete blood count)
* provide signed informed consent for study participation

Exclusion Criteria:

* history of allergies to melatonin products
* use of any drugs, vitamins, or supplements within 30 days before participation
* smoke or alcohol consumption within 1 week before participation
* blood or plasma donation within 30 days before participation

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-08 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Concentration-time profile after 2.5, 5, and 10 mg Melatonin niosomes (MN) oral gel single dose administration | 0, 15, 30, 45, 60, 75, 90, 120, 180, 240, 300, 360 and 480 min after MN oral gel administration
  Blood sampling

SECONDARY OUTCOMES:
Sleep induction effect (sleep onset latency, total sleep time, and wake after sleep onset) after 2.5, 5, and 10 mg MN oral gel single dose administration | 0-480 min after MN oral gel administration
  Sleep induction effect will be measured by using actigraph, behavior observation (all subjects), and Multiple sleep latency test (5 from 15 subjects).

OTHER OUTCOMES:
Adverse event after 2.5, 5, and 10 mg MN oral gel single dose administration | 0-24 h after MN oral gel administration
  nausea, vomiting, headache, irritability and others

CONTACTS AND LOCATIONS:
Overall Officials: Supawan Laohasiriwong, MD, Principal Investigator — Department of Otorhinolaryngology, Faculty of Medicine, Khon Kaen University
Locations (1):
- Academic Clinical Research Office, Amphur Muang, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Undecided